CLINICAL TRIAL: NCT00106249
Title: Treatment of Obsessive Compulsive Disorder (OCD) With Transcranial Magnetic Stimulation (TMS)
Brief Title: Transcranial Magnetic Stimulation (TMS) and Obsessive Compulsive Disorder (OCD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 5926R
Record Dates: First submitted 2005-03-21; First posted 2005-03-22 (Estimated); Results first posted 2017-01-27 (Estimated); Last update posted 2017-01-27 (Estimated); Status verified 2016-12

CONDITIONS: Obsessive-Compulsive Disorder
Keywords: TMS, Supplementary Motor Area, Obsessive-Compulsive Disorder
MeSH Terms: conditions — Obsessive-Compulsive Disorder | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Active rTMS (Active Comparator): Active Repetitive Transcranial Magnetic Stimulation (rTMS)
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation (rTMS)
- Sham rTMS (Sham Comparator): Placebo Repetitive Transcranial Magnetic Stimulation (rTMS)
  Interventions: Device: Sham

INTERVENTIONS:
Device: Repetitive Transcranial Magnetic Stimulation (rTMS) — Stimulus train of 30 min duration, 1Hz frequency, and 110% of the motor threshold intensity given once a day, 5 days a week, for 4 weeks by Magstim SuperRapid Magnetic Stimulator.
  Other Names: Magstim Rapid2, Magstim SuperRapid, Magstim Rapid, Magstim
  Arms: Active rTMS
Device: Sham — Sham rTMS will be administered using the Magstim Sham coil which contains a mu-metal shield that diverts the majority of the magnetic flux such that a minimal (less than 3%) magnetic field is delivered to the cortex in order to provoke a subjective sensation similar to that obtained with the real stimulation but without inducing significant cortical stimulation.
  Arms: Sham rTMS

SUMMARY:
This study will evaluate the clinical efficacy of functional Magnetic Resonance Imaging (fMRI) guided 1 Hz repetitive Transcranial Magnetic Stimulation (rTMS) applied to the Supplementary Motor Area (SMA) in OCD patients who have not fully responded to conventional therapies. The investigators will collect TMS measures of motor cortex excitability to test whether rTMS restores normal levels of intracortical inhibition found to be deficient in OCD. The investigators hypothesize that:

1. Compared to sham (placebo), active rTMS will improve symptoms of OCD as assessed with the Yale Brown Obsessive Compulsive Scale (Y-BOCS) and Clinical Global Impression (CGI).
2. Active (but not sham) rTMS will normalize levels of motor cortex excitability, as reflected by increased intracortical inhibition, motor threshold, and cortical silent period, and by decreased intracortical facilitation, relative to pre-treatment baseline.

DETAILED DESCRIPTION:
This study tests the efficacy of functional Magnetic Resonance Imaging (fMRI) guided repetitive Transcranial Magnetic Stimulation (rTMS) in the treatment of Obsessive Compulsive Disorder (OCD). This study also examines measures of brain function that may inform us about the brain basis underlying OCD.

Despite major advances in the study and treatment of OCD, patients often do not respond or experience only partial remission from pharmacotherapy or cognitive behavioral therapy. rTMS is a non-invasive procedure that allows stimulation of the brain using magnetic fields. Some studies have reported that rTMS may be helpful in reducing obsessive and compulsive symptoms. While promising, prior research has several limitations (e.g., relatively small sample sizes, stimulation of sub-optimal target areas, relatively short durations of treatment, and lack of sham (placebo) comparison).

This study addresses the drawbacks of prior work, and will provide data that will be important in determining whether rTMS can be useful for OCD patients resistant to conventional therapies. In this trial, 32 adult outpatients with OCD, that have been only partially responsive to conventional therapies, will be randomly assigned to one of two treatment groups (active low frequency (1 Hz) rTMS or sham-placebo) applied to the Supplementary Motor Area (SMA) daily for up to four weeks. If rTMS will be added onto ongoing pharmacotherapy, the doses must have been stable for 3 months prior to study entry. The SMA was selected because of its connections with areas of the brain, especially motor areas, implicated in OCD. Pilot work indicates that stimulation of SMA with low frequency rTMS was beneficial in OCD patients. Low frequency rTMS has the added benefit of a better safety profile (i.e. no risk of seizure) compared to high frequency rTMS.

Rating scales for symptom change will be obtained at baseline, during the rTMS course, and at the end of 4 weeks of treatment. Patients who do not meet response criteria after four weeks of sham and partial responders to either active or sham will be offered an open-label, cross-over phase for an additional four weeks of daily active rTMS treatment. Patients who meet response criteria in either the randomized phase or the cross-over phase will continue routine clinical care under the supervision of their treating psychiatrist, and will be invited back for a repeat assessment at 3 and 6 months to determine the persistence of benefit.

Measures of the excitability of the motor cortex have been reported to be abnormal in OCD, and may relate to dysfunction in motor pathways related to OCD circuits. We will collect measures of motor cortex excitability (performed with single pulse TMS) at baseline and after treatment to determine whether changes in these measures may be correlated with clinical improvement.

ELIGIBILITY:
Inclusion Criteria:

* Primary diagnosis of obsessive compulsive disorder, with residual OCD symptoms, defined as a total Y-BOCS score of ≥ 16, despite treatment with an adequate trial of a serotonin reuptake inhibitor (SRI), and a duration of the index episode of at least a year will be included. An adequate SRI trial is defined as treatment for at least 12 weeks on the SRI, that meets or exceeds the recommended dosage level for OCD (fluoxetine 60 mg/d, sertraline 200 mg/d, paroxetine 50 mg/d, fluvoxamine 250 mg/d, citalopram 60 mg/d, escitalopram 30 mg/d).
* Individuals who cannot tolerate medications of class and dose at the specified duration as described above will also be included.
* Patients currently on OCD medication must be at the same stable dose(s) and must continue to be under the care of their treating psychiatrist who will be writing prescriptions for concomitant medications through the duration of the study.

Exclusion Criteria:

* Refractory patients, where treatment refractoriness is defined as non-response to Clomipramine, at least 2 SSRIs at adequate dose and duration plus cognitive behavior therapy in the last year, will be excluded. An adequate trial of cognitive behavioral therapy is defined as at least once a week for 8 weeks with clear evidence of exposure during the sessions and homework given. Individuals diagnosed with major depressive disorder (current) of moderate or severe intensity (CGI ≥ 4), and those with bipolar disorder (lifetime), any psychotic disorder (lifetime), history of substance abuse or dependence within the past year (except nicotine and caffeine), and at significant acute suicide risk will also be excluded.

Other exclusion criteria include those common to every TMS protocol:

* Individuals with a clinically defined neurological disorder, with an increased risk of seizure for any reason, with a history of treatment with TMS, deep brain stimulation for any disorder will be excluded.
* Patients with cardiac pacemakers, implanted medication pumps, intracardiac lines, or acute, unstable cardiac disease, with intracranial implants (e.g. aneurysm clips, shunts, stimulators, cochlear implants, or electrodes) or any other metal object within or near the head, excluding the mouth, that cannot be safely removed will be excluded.
* Current use of any investigational drug will not be permitted.
* If participating in psychotherapy, patients must have been in stable treatment for at least three months prior to entry into the study, with no anticipation of change in frequency therapeutic sessions, or the therapeutic focus over the duration of the TMS trial.
* Finally, current significant laboratory abnormality, known or suspected pregnancy, women who are breast-feeding or women of childbearing potential not using a medically accepted form of contraception when engaging in sexual intercourse will also be excluded.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2004-11; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Mantovani, MD, PhD, Principal Investigator — Columbia University
Locations (1):
- New York State Psychiatric Institute, Experimental Therapeutics, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Maeda F, Pascual-Leone A. Transcranial magnetic stimulation: studying motor neurophysiology of psychiatric disorders. Psychopharmacology (Berl). 2003 Aug;168(4):359-76. doi: 10.1007/s00213-002-1216-x. Epub 2003 Jun 26. PMID 12830365
- [Background] Burt T, Lisanby SH, Sackeim HA. Neuropsychiatric applications of transcranial magnetic stimulation: a meta analysis. Int J Neuropsychopharmacol. 2002 Mar;5(1):73-103. doi: 10.1017/S1461145702002791. PMID 12057034
- [Background] Rossi S, Bartalini S, Ulivelli M, Mantovani A, Di Muro A, Goracci A, Castrogiovanni P, Battistini N, Passero S. Hypofunctioning of sensory gating mechanisms in patients with obsessive-compulsive disorder. Biol Psychiatry. 2005 Jan 1;57(1):16-20. doi: 10.1016/j.biopsych.2004.09.023. PMID 15607295
- [Background] Mantovani A, Simpson HB, Fallon BA, Rossi S, Lisanby SH. Randomized sham-controlled trial of repetitive transcranial magnetic stimulation in treatment-resistant obsessive-compulsive disorder. Int J Neuropsychopharmacol. 2010 Mar;13(2):217-27. doi: 10.1017/S1461145709990435. Epub 2009 Aug 20. PMID 19691873
- [Background] Mantovani A, Westin G, Hirsch J, Lisanby SH. Functional magnetic resonance imaging guided transcranial magnetic stimulation in obsessive-compulsive disorder. Biol Psychiatry. 2010 Apr 1;67(7):e39-40. doi: 10.1016/j.biopsych.2009.08.009. Epub 2009 Sep 30. No abstract available. PMID 19793582
- [Background] Mantovani A, Lisanby SH, Pieraccini F, Ulivelli M, Castrogiovanni P, Rossi S. Repetitive transcranial magnetic stimulation (rTMS) in the treatment of obsessive-compulsive disorder (OCD) and Tourette's syndrome (TS). Int J Neuropsychopharmacol. 2006 Feb;9(1):95-100. doi: 10.1017/S1461145705005729. Epub 2005 Jun 28. PMID 15982444

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Active rTMS | Sham rTMS
Started | 14 | 13
Completed | 11 | 11
Not Completed | 3 | 2
Not completed — Lost to Follow-up | 3 | 2

BASELINE CHARACTERISTICS:
Population: A total of 22 patients with at least 1 follow up were included in the final analyses. Four subjects only had baseline measure. The reason for them to withdraw from the study was their inability to attend daily treatment sessions due to schedule conflict with their job and long commute to the TMS laboratory.
Groups:
- Total: Total of all reporting groups
Arm/Group | Active rTMS | Sham rTMS | Total
Number analyzed (Participants) | 14 | 13 | 27
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.1 (13.1) | 37.1 (11.8) | 38.6 (12.5)
Gender [Count of Participants; unit: Participants]
  Female | 5 | 5 | 10
  Male | 9 | 8 | 17
Region of Enrollment [Number; unit: participants]
  United States | 14 | 13 | 27

OUTCOME MEASURES:

1. Primary Outcome: Clinical Improvement (Yale-Brown Obsessive Compulsive Scale/Y-BOCS)
Description: Response rate was defined as a decrease >25% on the YBOCS-SR. Y-BOCS-Self Report (Baer et al. 1993) is very similar to the clinician-administered one, and has shown excellent internal consistency and test-retest reliability, performing somewhat better than the interview (Steketee et al., 1996); subjects are asked to focus on the main obsessions and main compulsions and to answer five questions: time spent, interference, distress, resistance, and control. Consistent with the interview format, subjects rate each item on a 0 (none) to 4 (extreme) scale.
Time Frame: Through study completion
Measure: Number; unit: percentage of participants
Arm/Group | Active rTMS | Sham rTMS
Number analyzed (Participants) | 11 | 11
percentage of participants | 36 | 9
Statistical Analysis 1: Comparison: Active rTMS vs Sham rTMS; Test type: Superiority or Other; p < 0.05, ANOVA

2. Secondary Outcome: Motor Cortex Excitability (Motor Threshold)
Description: In 22 OCD patients, who completed the RCT, we applied the new customized software for acquisition and analysis of neurophysiology data that was developed to allow for automatic control of the TMS devices during motor cortex excitability measures. Specifically, the software delivers TMS pulses and automatically determines motor threshold (MT); a descending staircase method is utilized, starting at the intensity at which the optimal site selection for the MT is determined. After each stimulus in the MT experiments, the software would prompt the user to confirm the automated MEP-detection.
Time Frame: Through study completion
Population: repeated measure ANOVA, time X group interaction, right hemisphere MT
Measure: Mean (Full Range); unit: % MT change on right hemisphere
Arm/Group | Active rTMS | Sham rTMS
Number analyzed (Participants) | 11 | 11
% MT change on right hemisphere | 13 [0 to 100] | 0 [0 to 100]
Statistical Analysis 1: Comparison: Active rTMS vs Sham rTMS; Test type: Superiority or Other; p < 0.05, t-test, 2 sided

3. Secondary Outcome: Motor Cortex Excitability (Short Intracortical Inhibition)
Description: In 22 OCD patients enrolled in the RCT, we applied the new customized software for acquisition and analysis of neurophysiology data that was developed to allow for automatic control of the TMS devices during motor cortex excitability measures. For the paired-pulse (PP) measurements of short intracortical inhibition (SICI) the interstimulus interval (ISI) was set to 8-12 seconds on a continuous uniform distribution. The FPGA board samples the EMG data, controls the timing of the TMS stimuli, and also controls the intensity of the devices.
Time Frame: Through study completion
Population: Independent sample t-test, right hemisphere SICI
Measure: Mean (Full Range); unit: % change in conditioned/control MEP
Arm/Group | Active rTMS | Sham rTMS
Number analyzed (Participants) | 11 | 11
% change in conditioned/control MEP | 2.5 [0 to 3] | 1 [0 to 3]

ADVERSE EVENTS:
Arm/Group | Active rTMS | Sham rTMS
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/11
Other Adverse Events (participants affected / at risk) | 0/11 | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes